CLINICAL TRIAL: NCT02962947
Title: Melablock: A Multicentre Randomized, Double---blinded and Placebo---controlled Clinical Trial on the Efficacy and Safety of Once Daily Propranolol 80 mg Retard for the Prevention of Cutaneous Malignant Melanoma Recurrence
Brief Title: MELABLOCK: A Clinical Trial on the Efficacy and Safety of Propranolol 80 mg in Melanoma Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria di Firenze (Other)
Responsible Party: Principal Investigator, VINCENZO DE GIORGI, MD, MD, Azienda Sanitaria di Firenze
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT 2014---003970---18
Record Dates: First submitted 2016-02-19; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: Melanoma; Propanolol; Betablockers
MeSH Terms: conditions — Melanoma | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLACEBO (Placebo Comparator): Placebo will be taken daily during the study period
  Interventions: Drug: Placebo
- PROPRANOLOL (Active Comparator): Study participants in the treated group will take 80 mgR propranolol once daily .
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — 80 mgR propranolol once daily
  Arms: PROPRANOLOL
Drug: Placebo — placebo once daily
  Arms: PLACEBO

SUMMARY:
The effectiveness of propranolol in infantile hemangiomas, the apparent better response to propranolol in breast cancer and the use of propranolol in a proportion of patients who did not develop melanoma recurrence suggested to use this unselective β---blocker to test the study hypothesis. The investigators propose a randomized double---blind placebo---controlled clinical trial (RTC) to evaluate whether the treatment with propranolol 80 mgR/die reduce the risk of CMM recurrence and mortality. Patients with resected stage II/IIIA CMM will be recruited in various Centers in Italy. Participants will be randomly assigned to propranolol treatment or placebo (1:1 ratio), treated for at least 1 year and followed for 2 years. Recruitment will proceed simultaneously at the different Centers, and will be completed in 2 years. The primary outcome of the entire trial will be, however, estimated by assessing a reduction in overall mortality at five years. The investigators will also evaluate general CMM recurrence and CMM specific mortality.

DETAILED DESCRIPTION:
Cutaneous malignant melanoma (CMM) represents a major public health problem.Although melanoma accounts for only 4% of all dermatologic cancers, it is responsible for 80% of deaths from skin cancer; only 14% of patients with metastatic melanoma survive for five years . The probability of survival for melanoma stage II/IIIA at 15 years is around 50%.

Treatment with dacarbazine, fotemustine, temozolomide, interferon---α and interleukin---2 has been proposed in metastatic melanoma, but these drugs exert poor efficacy. More recently, ipilimumab, which blocks cytotoxic T---lymphocyte-associated antigen 4 to potentiate an antitumor T---cell response has been approved for the treatment of HLA---A*0201-positive patients with unresectable stage III or IV melanoma . This treatment has been found to delay mortality by about 4 months, although, in clinical trials a fraction of patients lived much longer . However, the drug caused severe or fatal side effects in almost 13% of patients, prompting the FDA to qualify its approval with a mitigation strategy. There were 14 deaths related to the study drugs (2.1%), and 7 were associated with immune---related adverse events. These findings do not suggest the use of ipilimumab in non metastatic patients. After surgical resection no specific pharmacotherapy is recommended for patients with stage II/IIIA CMM until metastases are found.

β---adrenoceptor antagonists (β---blockers) belong to one of the most widely used classes of drugs in clinical practice. Their use is mainly directed to the chronic management of hypertension , although they are also prescribed for ischemic heart disease, heart failure, anxiety, tremor, migraine and glaucoma , Initial pharmacoepidemiological evidence shows that β---blockers may reduce cancer risk. Indeed, β--- blockers have been reported to exert a certain degree of protection against prostate cancer . More recently, β---blocker treatment for concomitant diseases has been found to significantly reduce distant metastases, cancer recurrence, and cancer---specific mortality in breast cancer patients .

Infantile hemangiomas are the most common benign tumor of infancy. Over the last few years, propranolol has become a popular and successful treatment for infantile hemangiomas. The ability of ß---adrenoceptors to increase the vascular endothelial growth factor (VEGF) and the subsequent angionenetic pathway has contributed to the identification of this mechanism as a primary target of ß---blockers to limit cancer progression and to treat hemangiomas. The recent observation that propranolol treated successfully a case of infantile lymphangiomatosis and simulatneously reduced VEGF levels further strengthens this hypothesis. Preclinical studies have proposed that activation of β--- adrenoceptors play a detrimental role in melanoma, as in vitro studies showed that melanoma tissues expressed both β1--- and β2---adrenoceptors and that isoproterenol is a potent inducer of VEGF, IL---8 and IL---6 gene expression in human melanoma cells supporting the role of β--- adrenoceptors in this pathway. Thus, the role of ß---adrenoceptors to promote angiogenesis, supported by both basic and clinical evidence, represents the most robust working hypothesis explaining the beneficial effect of ß-blockers indifferent models of cancers,including melanoma.

In a prospective cohort of 121 consecutive patients with thick melanoma (Breslow >1), the investigators recently found that the use of β---blockers for concomitant diseases for 1 year or more is associated with a reduced risk of CMM recurrence. After a median follow---up time of 2.5 years, tumor progression was observed in 3.3% of the treated (n=30) subgroup and in 34.1% of the untreated (n=91) subgroup . Cox model on progression indicated a 36% (95%CI: 11%---54%; P=.002) risk reduction for each year of β---blocker use. No death was observed in the treated group, whereas in the untreated group 24 patients died. This study suggested for the first time that exposure to β---blockers is associated with a reduced risk of progression of thick CMM. In a larger group of 741 patients with thick and thin CMM the invetigators have recently confirmed the association between β---blocker prescription (79 patients) and the reduction in the risk of CMM recurrence and death.

The investigators hypothesize that treatment with propranolol reduces the risk of recurrence of CMM and decrease overall mortality.

Study Design The investigators propose a randomized double---blind placebo---controlled clinical trial (RTC) to evaluate whether the treatment with propranolol 80 mgR/die reduce the risk of CMM recurrence and mortality. Patients with resected stage II/IIIA CMM will be recruited in various Centers in Italy. Participants will be randomly assigned to propranolol treatment or placebo (1:1 ratio), treated for at least 1 year and followed for 2 years. Recruitment will proceed simultaneously at the different Centers, and will be completed in 2 years. Complete physical examination, measure of study compliance will be performed at baseline, as well as at the interim visits, every 4 months. The primary outcome of the entire trial will be, however, estimated by assessing a reduction in overall mortality at five years. The invetigators will also evaluate general CMM recurrence and CMM specific mortality.

Study population/Study Sites The proposed RCT will be conducted across Dermatology and Plastic Surgery centers primarily in Tuscany and also in other sites in Italy and if necessary in additional European countries. The end of follow-up is determined by recurrence, death, or last day of the follow-up.

Recruitment, Randomization and Treatment Assignment Potential study participants will be recruited among patients treated at Dermatology and Plastic Surgery centers in Tuscany/Italy. All screened subjects at each center will be assigned an ID number irrespective of whether or not they are randomized to receive study treatment. Randomization will be performed using a web---based procedure. Randomization patient numbers for each participant will be generated by computer for each of the two treatment assignments.

Unblinding will be provided once recruitment, data collection, laboratory analyses and whole follow up are completed. Protection of confidentiality will be achieved by limited access to the databases. At baseline the invetigators will also measure anthropometric variables such as weight, height. Arterial blood pressure, pulse rate and ECG will be recorded. Subjects enrolled will be asked about: hormone therapies, statin use; medical conditions such as xeroderma pigmentosum, basal cell nevus syndrome, lupus erythematosus, organ transplantation and immunosuppressive therapy; history of psoriasis; history of depression; all concomitant medications.

The participants will be asked to return to the recruitment clinic for 13 follow---up visits at months 4, 8, 12, 16, 20, 24, 28, 32, 36, 42, 48, 54 and 60. At alternate visits they will receive the next 8 months supply of medication for the study participants. The physician will perform a complete physical examination, including measurement of body weight, blood pressure and pulse rate, to assess the general health of the study participant. We will collect up---dated information about health status and signs of recurrence of melanoma.

Dosage and Administration Study participants will be randomized to 80 mgR propranolol once daily or placebo.

Concomitant medications Patients will be discouraged from taking unspecified medications. However all medications, vitamin and mineral supplements and herbs taken by the participant should be documented on the Case Report Form (CRF) and will include: start and stop date, dose and route of administration, and indication for use.

Methods to monitor adherence The following methods of adherence monitoring will be used: blisters evaluation and subject self--- reporting, in keeping with the current practice of investigators to rely heavily on such tools.

Withdrawal criteria Study Participants will be able to withdraw from the study at any time. Reason for subject discontinuation may include: recurrence, adverse event that compromises the patient's ability to participate in the study, such as serious acute emergencies (i.e., heart attack, stroke or acute abdomen surgery). Subjects who discontinue treatment will be encouraged to participate in the follow---up examinations to maintain an intention---to---treat analysis.

After 3 years of treatment patients will terminate the intervention period and will be followed on an annual basis for 2 years unless the early termination of the study. After 546 patients have been randomized, the accrual will be closed. When the last randomized subject has concluded the 3 years of treatment and 2 years of follow---up, the study will be considered closed. The Data Safety and Monitoring Board (DSMB), the Ethics Committee and regulatory authorities can make the decision to terminate the study earlier. This decision could be based on factors such as unacceptable adverse events, poor accrual or compliance on interim analyses.

Staffing and Scheduling Coordinating Centre for Field Activities: the study will have a study coordination center at the Department of Preclinical and Clinical Pharmacology of the University of Florence, which will coordinate all the different aspects of the study field conduction. Prof. Alessandro Mugelli expert in cardiopharmacology, Prof. Niccolò Marchionni, expert in clinical cardiology and Dr. Sara Gandini, expert in data management and biostatistics will assist Dr. Vincenzo De Giorgi and Prof. Pierangelo Geppetti in the coordination of the study. The clinical investigators led by the PI, Dr. Vincenzo De Giorgi, will be responsible for study recruitment, clinical examination of patients and assessing patient safety. Study set-up will take approximately 6 months and will occur at the beginning of the funding period. After 6 months of study set---up period and 9 years of active data collection period (i.e., time between the first person entering the trial up to the last person completing the final 24 month follow-up visit), the last 6 months will be for study close---out activities. These activities will include final data entry and cleaning, final data analysis, and report writing. The entire study from beginning of study set-up to end of study close-out will take 7 years to be completed (two years of accrual, 3 years of treatment, 2 years of follow-up).

Sample size calculations Results of the previous prospective study on of 741 melanoma patients showed that, after a median follow---up time of 4 years, Cox-regression model on overall mortality indicated a 38% (95%CI: 10%---57%;P=.02) risk reduction for each year of β--blocker use. Cautiously, we considered an hazard ratio of about 0.6 for the randomized placebo-controlled phase-II trial. A total sample size of 546 (split equally between the two groups) will give us 90% of power for estimating a improvement in OS at five years achieves 90% power to detect an improvement given a survival at five years of 0.70 and an increase to 0.82 in the treatment groups)at a significance level (alpha) of 0.05 using a two---sided log rank test. These results assume that 3 sequential tests are made using the O'Brien-Fleming spending function to determine the test boundaries and that the hazards are proportional.

ELIGIBILITY:
Inclusion Criteria:

1. Stage: Ib (T1b, T2a), IIa (T2b, T3a), IIb (T3b T4a) and IIc (T4b), N0, M0; IIIA (N1a, N1b)
2. Signed Informed Consent;
3. Performance Status of 0---1 (ECOG);
4. Hematopoietic functionality at the entry of the study: leukocytes, platelets, hemoglobin and neutrophils within the normal limits of laboratory references;
5. Hepatic and renal functionality at the entry of the study: LDH, bilirubin, AST, ALT, alkalinephosphatase, BUN and serum creatinine within the normal range of each laboratory;

Exclusion Criteria:

1. Primary not cutaneous melanoma;
2. Clinical/radiological evidence or laboratory/pathology report of not completely resectedmelanoma;
3. History of cancer
4. Current use or past use in the last two years of any b---blockers for any other medical condition
5. Current use of verapamil, diltiazem or similar calcium channel blocker
6. Current use of centrally acting antihypertensive drugs as α---methyldopa, clonidine
7. Hypersensitivity to propranolol or to any of the excipients;
8. Acute heart failure or during episodes of heart failure decompensation requiring i.v.

   inotropic therapy;
9. Cardiogenic shock;
10. Sinoatrial block ;
11. Second or third degree atrio---ventricular block;
12. Marked bradycardia (less than 60 beats/min) ;
13. Extreme hypotension (systolic blood pressure <100mmHg) ;
14. Severe asthma or severe chronic obstructive pulmonary disease ;
15. Sick sinus syndrome;
16. Severe forms of peripheral arterial occlusive disease and Raynaud's syndrome;
17. Metabolic acidosis
18. Asthma
19. Diabetes
20. Heart failure
21. History of psoriasis
22. Pregnancy or breast feeding or planning on becoming pregnant during the 3 years of treatment (for major details see the Section "Pregnancy in the Study", below);
23. Any medical condition that in the physician's opinion would potentially interfere with the patient ability to adhere to protocol and treatment;
24. Any logistic condition that do not allow follow---up of the disease of the patient.
25. Hypersensitivity to propranolol, child bearing or breastfeeding.
26. Pheocromocytoma 27. Prinzmetal's Angina 28. Fasting -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2017-06; Primary Completion 2019-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Effect of Propranolol on overall survival for melanoma patients in stage II/IIIA (T2, N0 or N1, M0) | 5 years
  To assess the effect of treatment with propranolol 80 mg retard (R) on overall survival for cutaneous malignant melanoma (CMM) patients in stage II/IIIA (T2, N0 or N1, M0) at five years of follow---up,after at least one year of treatment. Chi-square and Fisher's exact tests will be used to analyze the associations between the categorical variables. Logistic regression adjusting for confounding factors will be also performed. Wilcoxon tests will be used to compare continuous variables. Overall survival and Disease Free Survival curves will be estimated by the Kaplan-Meier method. Log-rank test will be used to compare survival time between groups and Cox proportional hazards models to evaluate the effect of β-blockers treatment and duration of treatment on melanoma recurrence and mortality, considering stratification factors.

SECONDARY OUTCOMES:
Effect of Propranolol on disease free survival for melanoma patients in stage II/IIIA | 5 years
  To evaluate the effect of treatment on disease free survival (DFS) at five years for CMM patients in stage II/IIIA. Chi-square and Fisher's exact tests will be used to analyze the associations between the categorical variables. Logistic regression adjusting for confounding factors will be also performed. Wilcoxon tests will be used to compare continuous variables. Overall survival and Disease Free Survival curves will be estimated by the Kaplan-Meier method. Log-rank test will be used to compare survival time between groups and Cox proportional hazards models to evaluate the effect of β-blockers treatment and duration of treatment on melanoma recurrence and mortality, considering stratification factors.
Effect of propranolol on specific mortality for melanoma patients in stage II/IIIA | 5 years
  To evaluate the effect of treatment on specific mortality for CMM patients in stage II/IIIA. Chi-square and Fisher's exact tests will be used to analyze the associations between the categorical variables. Logistic regression adjusting for confounding factors will be also performed. Wilcoxon tests will be used to compare continuous variables. Overall survival and Disease Free Survival curves will be estimated by the Kaplan-Meier method. Log-rank test will be used to compare survival time between groups and Cox proportional hazards models to evaluate the effect of β-blockers treatment and duration of treatment on melanoma recurrence and mortality, considering stratification factors.
Effect of propranolol treatment on the long-term safety on melanoma patients in stage II/IIIA | 5 years
  To evaluate the long---term safety of treatment on CMM patients in stage II/IIIA.This study will use the NCI Common Terminology Criteria for Adverse events version 3.0, for toxicity and adverse event reporting. The CTCAE provides descriptive terminology and a grading scale for each adverse event listed. A copy of the CTCAE can be found at http://ctep.cancer.gov. AEs will be assessed according to the CTCAE grade associated with the AE term. AEs that do not have a corresponding CTCAE term will be assessed according to their impact on the participant's ability to perform daily activities

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronow WS. Current role of beta-blockers in the treatment of hypertension. Expert Opin Pharmacother. 2010 Nov;11(16):2599-607. doi: 10.1517/14656566.2010.482561. Epub 2010 Apr 28. PMID 20426702
- [Background] Barron TI, Connolly RM, Sharp L, Bennett K, Visvanathan K. Beta blockers and breast cancer mortality: a population- based study. J Clin Oncol. 2011 Jul 1;29(19):2635-44. doi: 10.1200/JCO.2010.33.5422. Epub 2011 May 31. PMID 21632503
- [Background] Bielecka-Dabrowa A, Aronow WS, Rysz J, Banach M. Current place of beta-blockers in the treatment of hypertension. Curr Vasc Pharmacol. 2010 Nov;8(6):733-41. doi: 10.2174/157016110793563861. PMID 20626337
- [Background] Chen JM, Heran BS, Perez MI, Wright JM. Blood pressure lowering efficacy of beta-blockers as second-line therapy for primary hypertension. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD007185. doi: 10.1002/14651858.CD007185.pub2. PMID 20091622
- [Background] Cruickshank JM. Are we misunderstanding beta-blockers. Int J Cardiol. 2007 Aug 9;120(1):10-27. doi: 10.1016/j.ijcard.2007.01.069. Epub 2007 Apr 12. PMID 17433471
- [Background] De Giorgi V, Gandini S, Grazzini M, Benemei S, Marchionni N, Geppetti P. Effect of beta-blockers and other antihypertensive drugs on the risk of melanoma recurrence and death. Mayo Clin Proc. 2013 Nov;88(11):1196-203. doi: 10.1016/j.mayocp.2013.09.001. PMID 24182700
- [Background] De Giorgi V, Grazzini M, Gandini S, Benemei S, Lotti T, Marchionni N, Geppetti P. Treatment with beta-blockers and reduced disease progression in patients with thick melanoma. Arch Intern Med. 2011 Apr 25;171(8):779-81. doi: 10.1001/archinternmed.2011.131. PMID 21518948
- [Background] Lamy S, Lachambre MP, Lord-Dufour S, Beliveau R. Propranolol suppresses angiogenesis in vitro: inhibition of proliferation, migration, and differentiation of endothelial cells. Vascul Pharmacol. 2010 Nov-Dec;53(5-6):200-8. doi: 10.1016/j.vph.2010.08.002. Epub 2010 Aug 20. PMID 20732454
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Lemeshow S, Sorensen HT, Phillips G, Yang EV, Antonsen S, Riis AH, Lesinski GB, Jackson R, Glaser R. beta-Blockers and survival among Danish patients with malignant melanoma: a population-based cohort study. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):2273-9. doi: 10.1158/1055-9965.EPI-11-0249. Epub 2011 Sep 20. PMID 21933972
- [Background] Lyons KE, Pahwa R. Pharmacotherapy of essential tremor : an overview of existing and upcoming agents. CNS Drugs. 2008;22(12):1037-45. doi: 10.2165/0023210-200822120-00006. PMID 18998741
- [Background] Miller AJ, Mihm MC Jr. Melanoma. N Engl J Med. 2006 Jul 6;355(1):51-65. doi: 10.1056/NEJMra052166. No abstract available. PMID 16822996
- [Background] Ozeki M, Fukao T, Kondo N. Propranolol for intractable diffuse lymphangiomatosis. N Engl J Med. 2011 Apr 7;364(14):1380-2. doi: 10.1056/NEJMc1013217. No abstract available. PMID 21470038
- [Background] Perron L, Bairati I, Harel F, Meyer F. Antihypertensive drug use and the risk of prostate cancer (Canada). Cancer Causes Control. 2004 Aug;15(6):535-41. doi: 10.1023/B:CACO.0000036152.58271.5e. PMID 15280632
- [Background] Tsao H, Atkins MB, Sober AJ. Management of cutaneous melanoma. N Engl J Med. 2004 Sep 2;351(10):998-1012. doi: 10.1056/NEJMra041245. No abstract available. PMID 15342808
- [Background] Williams B. Beta-blockers and the treatment of hypertension. J Hypertens. 2007 Jul;25(7):1351-3. doi: 10.1097/HJH.0b013e328182266a. No abstract available. PMID 17563554
- [Background] Wiysonge CS, Bradley H, Mayosi BM, Maroney R, Mbewu A, Opie LH, Volmink J. Beta-blockers for hypertension. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD002003. doi: 10.1002/14651858.CD002003.pub2. PMID 17253471